CLINICAL TRIAL: NCT03744832
Title: Point of Care Group A Streptococcal Testing in a Pediatric Emergency Department: A Randomized Controlled Trial
Brief Title: Point of Care Streptococcal Pharyngitis Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Quynh Doan, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H18-02371
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Pharyngitis Acute
Keywords: Pediatrics; Emergency Department; Point of Care Testing; Group A Strep
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point of Care Testing (Experimental): Point of care testing using the Alere i™ Strep A assay for patients randomized to this study arm when presenting with suspected streptococcal pharyngitis and having their throat swabbed. If test is positive, patients will be started on antibiotics prior to discharge from the ED. If test is negative, patients will not be started on antibiotics.
  At home, the patient family will be asked to complete an online survey and/or keep a written diary daily detailing their clinical course following discharge from the ED.
  Interventions: Diagnostic Test: Alere i™ Strep A assay
- Standard Care (Active Comparator): Conventional testing using a standard bacterial throat culture for patients randomized to this study arm when presenting with suspected streptococcal pharyngitis and having their throat swabbed. Patients will be discharged with a post-dated prescription and will be contacted in approximately 3 days if their culture results are positive to fill/take the antibiotics.
  At home, the patient family will be asked to complete an online survey and/or keep a written diary daily detailing their clinical course following discharge from the ED.
  Interventions: Diagnostic Test: Throat culture

INTERVENTIONS:
Diagnostic Test: Alere i™ Strep A assay — Point of care (POC) molecular-based, nucleic acid amplification test (NAAT). This isothermal molecular assay is CLIA waived (Clinical Laboratory Improvement Amendments) and Health Canada licensed for POC use, and is anticipated to have approval for use without need for back up culture testing.
  Arms: Point of Care Testing
Diagnostic Test: Throat culture — Standard bacterial throat culture.
  Arms: Standard Care

SUMMARY:
Sore throat is a common problem in children typically caused by viral or bacterial infections. While viral infections resolve without treatment, bacterial infections, such as "strep throat," are treatable with antibiotics. Diagnosing "strep throat" traditionally required a throat swab for culture that delays treatment for several days. This may result in prolonged illness, activity absenteeism, and significant healthcare costs. New molecular tests can accurately diagnose "strep throat" within 8 minutes, but are more expensive and require impact evaluation before widespread implementation. This study will compare a new bedside molecular test with conventional throat cultures to evaluate for benefits to patients and families seen in the emergency department, as well to healthcare system operations. The investigators hypothesize that care for children and the associated healthcare costs will improve with these point of care molecular tests.

DETAILED DESCRIPTION:
Purpose:

Molecular-based, nucleic acid amplification tests (NAATs), have been proposed as a diagnostic solution for streptococcal pharyngitis. Indeed, available data suggest that NAATs have similar performance to conventional culture testing, and point of care (POC) NAATs recently became commercially available. These bedside tests do not require operation by laboratory personnel and have been approved by Health Canada for use without the need for backup culture testing. This study seeks to compare the clinical outcomes of a POC NAAT approach with a conventional bacterial culture-based approach for children presenting to a Pediatric Emergency Department (PED) with suspected streptococcal pharyngitis. Results from this clinical trial will elicit critical information regarding the potential clinical benefit of implementing this new technology in the PED.

Hypothesis:

The investigators hypothesize that clinical outcomes (duration of illness, incidence of complications, absenteeism) and system utilization (PED length of stay, ancillary testing, return visits to hospital or community healthcare facility, appropriate antibiotic treatment) will improve with a POC NAAT diagnostic approach for suspected streptococcal pharyngitis.

Justification:

Determining the etiology of pharyngitis is necessary, both to minimize inappropriate antimicrobial therapy for viral infections, and to reduce the incidence of complications, duration of illness, and transmission of streptococcal infections, for which antibiotics are indicated. However, signs and symptoms of viral and streptococcal pharyngitis overlap significantly, and accurate differentiation based on history and clinical examination is difficult even for experienced clinicians. As a result, the Infectious Diseases Society of America (IDSA) currently recommends swabbing the throat and testing for streptococcal pharyngitis by culture, which is the current standard of practice at BC Children's Hospital (BCCH). However, while bacterial cultures are accurate and economical, they are often clinically impractical and cause delay in treatment due to the relatively long lag time (>48 hours) between collection of the specimen and final microbiological diagnosis. Available data suggest that new POC NAATs have similar performance to conventional culture testing with results available within 8 minutes. This could potentially improve clinical outcomes and reduce system utilization, but implementation would require significant task shifting, logistical support, and additional training. This study will provide an impact evaluation of this new technology in a PED, which is a necessary first step prior to implementation, in an effort to ultimately improve care for children and youth while minimizing costs to society.

Objectives:

The primary objective of this study is to compare POC NAAT testing with conventional throat culture testing (the current standard of care) for children and adolescents presenting to a PED for suspected streptococcal pharyngitis with regards to clinical management, symptom resolution, and resource utilization.

Demographic and Visit Characteristics:

1. Age in years
2. Sex (Male or Female)
3. Triage acuity level using the Canadian Triage and Acuity Scale (CTAS)
4. Visit day of the week (weekday/weekend/holiday)
5. Length of stay (minutes) using date and time of arrival (registration/triage) and date and time of discharge
6. McIsaac score (0-5)
7. Disposition

Statistical Analysis:

Descriptive statistics will be used to summarize study population demographic and baseline characteristics. The Student t-test will be applied for continuous variables (mean time to symptom resolution, mean days off, etc.), and the chi-square test will be applied for categorical variables (proportion appropriately treated).

Quality Assurance:

Left over swabs from either study arm will be stored to subsequently culture or conduct NAAT testing for patients randomized to the interventional (POC testing) or standard (conventional culture) study arms, respectively. This alternate method testing will not be conducted until the end of the study, unless culture and sensitivity testing is required earlier for a patient that is randomized to the interventional POC study arm with a known severe beta-lactam allergy and/or does not respond to second-line therapy. The POC test performance will not be evaluated as part of this study as it has been determined to be at least equivalent to culture detection in the past.

Sample size estimation:

Using published literature on the effect of antibiotics on GAS pharyngitis, we estimate that the mean time to resolution in the POC group is 3 days (with a standard deviation of 2 days), and a minimally important difference in mean time to resolution between the groups being 1.5 days. Using 80% power at a significance level of 0.05, the required sample size is 28 subjects per group. With an estimated 30% positivity rate, and accounting for 10% of individuals lost to follow-up, the investigators will aim to recruit 100 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-17 years of age who seek care in a ED with sore throat, and in whom the ED clinician is considering a throat swab for culture for suspected GAS pharyngitis. In addition, only English speaking families will be recruited.

Exclusion Criteria:

* Patients younger than 3 and older than 17 years of age will be excluded. In addition, patients who had a throat swab completed and/or were treated with antibiotics prior to presenting to the ED for the current illness, and patients with underlying cardiorespiratory illness will be excluded.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Sore throat resolution. | 7 days.
  Mean time in half-days from ED discharge to sore throat resolution (POC vs. standard).

SECONDARY OUTCOMES:
Fever resolution. | 7 days.
  Mean time in half-days from ED discharge to fever resolution (axillary temperature; POC vs. standard).
Appropriate antibiotic utilization by patients/families. | 7 days.
  Proportion of patients appropriately treated with antibiotics (ie. streptococcal-positive treated with antibiotics and streptococcal-negative not started on antibiotics. Families may decide to fill prescription without a positive culture result or families may obtain a prescription from elsewhere despite a negative POC test in the ED; POC vs. standard).
Calls averted. | 7 days.
  Number of patient calls averted (POC vs. standard).
Parental Absenteeism. | 7 days.
  Mean number of days away from work for a parent (measured by half day units; POC vs. standard).
Child Absenteeism | 7 days
  Mean number of days away from school/daycare for a child
Healthcare return visits. | 7 days.
  Proportion of patients with a least 1 ED re-visit or community healthcare facility visit for the same illness within 7 days (POC vs. standard).
Length of stay. | 7 days.
  length of stay (LOS) will be calculated from time of registration/triage until discharge (POC vs. standard).
Ancillary testing. | 7 days
  May include, but is not limited to, a complete blood count, urinalysis, urine culture, blood, culture, or neck/chest radiographs (POC vs. standard).

CONTACTS AND LOCATIONS:
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.

REFERENCES:
- [Derived] Gill C, Chui C, Goldfarb DM, Meckler G, Doan Q. Molecular Point-of-Care Testing in the Emergency Department for Group A Streptococcus Pharyngitis : A Randomized Trial. Pediatr Emerg Care. 2024 Sep 1;40(9):632-637. doi: 10.1097/PEC.0000000000003154. Epub 2024 Mar 18. PMID 38498934